CLINICAL TRIAL: NCT01911793
Title: Stoma Tube Decompression and Postoperative Ileus After Major Colorectal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough staff resource to complete study.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Director of Colorectal Surgery Residency, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Stoma Tube Study
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Ileus; Bowel Obstruction
Keywords: stoma; ileus; postoperative; stoma tube
MeSH Terms: conditions — Ileus; Intestinal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stoma tube (Experimental): Stoma tube (18 French) red robinson catheter inserted into stoma at the time of surgery
  Interventions: Device: Stoma Tube
- Standard Stoma (No Intervention): Patients will have standard stoma created without insertion of stoma tube. Stoma tube will only be inserted postoperative if the patient is felt to have postoperative ileus, nausea, vomiting, and decreased stoma output as per standard protocol.

INTERVENTIONS:
Device: Stoma Tube — Stoma tube will be inserted into stoma at the time of surgery for patients assigned to Stoma Tube group.
  Other Names: Red robinson catheter
  Arms: Stoma tube

SUMMARY:
Postoperative ileus is common after colorectal surgery, occurring in up to 20% of patients. Stomas are frequently created in conjunction with major colorectal surgery. Obstruction at the level of the stoma is a common cause of bowel obstruction or ileus. This is often manifested by decrease or delay in stoma output and is often attributed to edema at the level of the stoma. Thus, a temporary tube (red robinson catheter) is placed into the stoma at bedside, which often relieves the obstruction until the edema at the level of the stoma resolves and stoma function occurs around the temporary tube. At this time, the tube is removed and the stoma continues to function normally.

The purpose of this study is to evaluate whether a stoma tube (red-robinson catheter) placed at the time of stoma creation would reduce the incidence of postoperative ileus in patients undergoing major colorectal surgery with creation of a stoma.

ELIGIBILITY:
Inclusion Criteria:

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males or females, 18> years of age and older inclusive at the time of study screening;
3. American Society of Anesthesiologists (ASA) Class I-III (Appendix III);
4. Due to undergo ileostomy or colostomy creation via laparotomy or laparoscopy;

Exclusion Criteria:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures;
2. American Society of Anesthesiologists (ASA) Class IV or V;
3. Children <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Fleshner, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Iyer S, Saunders WB, Stemkowski S. Economic burden of postoperative ileus associated with colectomy in the United States. J Manag Care Pharm. 2009 Jul-Aug;15(6):485-94. doi: 10.18553/jmcp.2009.15.6.485. PMID 19610681
- [Background] Akesson O, Syk I, Lindmark G, Buchwald P. Morbidity related to defunctioning loop ileostomy in low anterior resection. Int J Colorectal Dis. 2012 Dec;27(12):1619-23. doi: 10.1007/s00384-012-1490-y. Epub 2012 May 11. PMID 22576906
- [Background] Le Q, Liou DZ, Murrell Z, Fleshner P. Does a history of postoperative ileus predispose to recurrent ileus after multistage ileal pouch-anal anastomosis? Tech Coloproctol. 2013 Aug;17(4):383-8. doi: 10.1007/s10151-012-0942-2. Epub 2012 Nov 27. PMID 23183687

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Stoma: Patients will have standard stoma created without insertion of stoma tube. Stoma tube will only be inserted postopertively if the patient is felt to have postopeprative ileus, nausea, vomiting, and decreased stoma output as per standard protocol.
Period: Overall Study
Arm/Group | Stoma Tube | Standard Stoma
Started | 1 | 5
Completed | 0 | 0
Not Completed | 1 | 5
Not completed — Physician Decision | 1 | 5

BASELINE CHARACTERISTICS:
Population: Data were not collected and no data was analyzed study was terminated due to issues with study enrollment and study administrative coverage.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stoma Tube | Standard Stoma | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Tolerating Low Residue Diet
Description: % of patients tolerating a low residue diet on postoperative day 3 will be assessed
Time Frame: by postoperative day 3( 3rd day after surgery)
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Flatus (Passing Gas Into Stoma Bag)
Description: # of hours after surgery at which point first passage of flatus (gas) into stoma bag
Time Frame: during 30 day postoperative period
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Passage of Stool
Description: # of hours after surgery until the patient passes stool into stoma bag
Time Frame: during 30 day postoperative period
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Discharge
Description: postoperative day after surgery which patient was discharged home
Time Frame: 30 day postoperative period
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Discharge Based on GI Function
Description: postoperative day which patient is considered ready for discharge based solely on Gastrointestinal function
Time Frame: 30 day postoperative period
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Major and Minor Medical and Surgical Complications
Description: any major or minor medical and surgical complications after surgery will be recorded
Time Frame: 30 day postoperative period
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Any Insertion of Nasogastric Tube
Description: insertion of nasogastric tube after surgery will be recorded
Time Frame: 30 day postoperative period
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Episodes of Vomiting
Description: any episodes of vomiting will be recorded
Time Frame: during postoperative hospital admission (30 day period)
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Diagnosis of Postoperative Ileus
Description: diagnosis of postoperative ileus or bowel obstruction made by attending surgeon based on clinical data including abdominal distention, nausea/vomiting, decreased stom output and radiologic factors
Time Frame: 30 day postoperative period
Population: as for baseline characteristics
Arm/Group | Stoma Tube | Standard Stoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data were not collected and no data was analyzed study was terminated due to issues with study enrollment and study administrative coverage. Total Number of Participants at Risk (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for this study.
Description: Data were not collected and no data was analyzed study was terminated due to issues with study enrollment and study administrative coverage.
  Total Number of Participants at Risk (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Stoma Tube | Standard Stoma
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study only accrued 6 patients. Due to poor enrollment and issues with administrative coverage for study it was decided to terminate the study.

NO data analysis has been done and will not be done in the future. This study was closed with the IRB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No